

## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

## **Study Information**

| Title Protocol number Protocol version identifier Date | Real-World Effectiveness of Tafamidis 80 mg or 61 mg on<br>Neurologic Disease Progression in Patients with Mixed-Phenotype<br>Variant Transthyretin Amyloid Cardiomyopathy (ATTRv-CM)<br>B3461099<br>v3.0 |
|---|---|
| Active substance | N07XX08 |
| Medicinal product | Tafamidis |
| Research question and objectives | Primary objective: • To assess neurologic function before and after initiation of tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, in patients with mixed-phenotype ATTRv-CM in a real-world setting Secondary objective: • To assess modified body mass index (mBMI) in patients with mixed-phenotype ATTRv-CM receiving tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, in a real-world setting |
| Author | PPD (Main Author) PPD |

## Tafamidis B3461099 NON-INTERVENTIONAL STUDY PROTOCOL Amendment 2, Version 3.0, 31 May 2023

| PPD |
|-----|

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

## 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 3 |
|---------------------------------------------------------------------|----|
| 2. LIST OF ABBREVIATIONS | 5 |
| 3. RESPONSIBLE PARTIES | 7 |
| 4. ABSTRACT | 7 |
| 5. AMENDMENTS AND UPDATES | 8 |
| 6. MILESTONES | 9 |
| 7. RATIONALE AND BACKGROUND | 9 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 11 |
| 9. RESEARCH METHODS | 11 |
| 9.1. Study Design | 11 |
| 9.2. Setting. | 12 |
| 9.2.1. Inclusion Criteria | 12 |
| 9.2.2. Exclusion Criteria | 12 |
| 9.3. Variables | 13 |
| 9.3.1. Exposure Variables | 13 |
| 9.3.2. Outcome Variable | 13 |
| 9.4. Data Source | 15 |
| 9.5. Study Size | 15 |
| 9.6. Data Management | 15 |
| 9.7. Data Analysis | 16 |
| 9.8. Quality Control | 16 |
| 9.9. Limitations of the Research Methods | 17 |
| 9.10. Other Aspects | 17 |
| 10. PROTECTION OF HUMAN SUBJECTS | 17 |
| 10.1. Patient Information | 17 |
| 10.2. Patient Consent | 18 |
| 10.3. Institutional Review Board (IRB)/Independent Ethics Committee | 18 |
| 10.4. Ethical Conduct of the Study | 18 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE | 10 |

## Tafamidis B3461099 NON-INTERVENTIONAL STUDY PROTOCOL Amendment 2, Version 3.0, 31 May 2023

| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 18 |
|-------------------------------------------------------------|----|
| 13. REFERENCES | 19 |
| 14. LIST OF TABLES | 21 |
| 15. LIST OF FIGURES | 21 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 21 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 21 |
| ANNEX 3. ADDITIONAL INFORMATION | 21 |

## 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ANOVA | Analysis of variance |
| ATTR-ACT | Transthyretin amyloidosis cardiomyopathy clinical trial |
| ATTR-CM | Transthyretin amyloid cardiomyopathy |
| ATTR-PN | Transthyretin amyloid polyneuropathy |
| ATTRv | Variant transthyretin amyloidosis |
| ATTRv-CM | Variant transthyretin amyloid cardiomyopathy |
| ATTRwt | Wild-type transthyretin amyloidosis |
| BMI | Body mass index |
| CCI | Charlson Comorbidity Index |
| CMTNS2 | Charcot-Marie-Tooth neuropathy score v2 |
| CI | Confidence interval |
| EMR | Electronic medical record |
| FTP | File transfer protocol |
| GPP | Good pharmacoepidemiology practices |
| HIV | Human immunodeficiency virus |
| ID | Identifier |
| IRB | Institutional review board |
| IP | Internet protocol |
| ISPOR | International Society for Pharmacoeconomics and<br>Outcomes Research |
| mBMI | Modified body mass index |
| NIS-CS | Neuropathy impairment score-composite score |
| NIS-LL | Neuropathy impairment score-lower limbs |
| MMRM | Mixed model repeated measures |
| MRC | Medical Research Council |
| PND | Polyneuropathy disability |
| REDCap | Research Electronic Data Capture |

| Abbreviation | Definition |
|--------------|-----------------------------|
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis System |
| SD | Standard deviation |
| TTR | Transthyretin |
| QA | Quality assurance |
| QC | Quality control |

## 3. RESPONSIBLE PARTIES

## Principal Investigator(s) of the Protocol

| Name, degree(s) | Job Title | Affiliation | Address |
|-----------------|-----------|-------------|---------|
| PPD | | | |

## Additional Responsible Parties for the Study

| Name, degree(s) | Job Title | Affiliation | Email Address |
|-----------------|-----------|-------------|---------------|
| PPD | | | |

## 4. ABSTRACT

Standalone document - Annex 1.

## 5. AMENDMENTS AND UPDATES

| Amendment<br>number | Date | Protocol<br>section(s)<br>changed | Summary of amendment(s) | Reason |
|---|---|---|---|---|
| Amendment<br>1 | 01/09/23 | 1-6, 9, 11 | Administrative amendment: Number and timing of measurements changed to address data availability. Addition of CMTNS2 instrument. Updated template language for data analysis Updated AE reporting language per SOP | Change in PIs and available data. Not expecting most patients to have multiple measures before or after treatment. |
| Amendment<br>2 | 31 May<br>2023 | Inclusion Criteria,<br>Section 9.21 | Changed criteria number 4 from "≥2: to "≥1" | Administrative, typographical error |
| Amendment<br>2 | 31 May<br>2023 | Table 9-2, Clinical<br>Outcomes | Deleted footnote to align with SAP | Administrative |

#### 6. MILESTONES

| Milestone | Planned date |
|--------------------------------------|------------------|
| Completion of feasibility assessment | 30 October 2022 |
| Start of data collection | 28 February 2023 |
| End of data collection | 01 November 2023 |
| Final study report | 01 October 2024 |

#### 7. RATIONALE AND BACKGROUND

ATTR amyloidosis is a progressive, life-threatening, and heterogeneous rare disease caused by the deposition of transthyretin-derived amyloid fibrils in the peripheral nerves, heart, and other organs. <sup>1,2</sup> ATTR amyloidosis may arise from variants (mutations) in the transthyretin (TTR) gene (ATTRv amyloidosis), with more than 140 ATTRv genotypes having been identified, <sup>3</sup> or from the aggregation of non-mutated wild-type TTR (ATTRwt amyloidosis). Amyloid deposition in the peripheral nerves results in transthyretin amyloid polyneuropathy (ATTR-PN), but multiple symptoms and system involvement are hallmarks of ATTR-PN. <sup>2,4,5</sup> Amyloid fibril deposition in the extracellular matrix of the heart <sup>2,6</sup> results in ATTR-CM, which is characterized by arrhythmias and heart failure. <sup>7,8</sup> ATTRwt amyloidosis predominantly manifests as ATTR-CM. ATTRv amyloidosis is now widely recognized as a spectrum of disease that can manifest as polyneuropathy, cardiomyopathy, or a mixed phenotype, depending on the particular TTR variant, amyloid deposition pattern, and multisystem involvement.

Tafamidis meglumine is a first-in-class highly specific and selective stabilizer of both wild-type and amyloidogenic variants of transthyretin (TTR)<sup>9</sup> developed for the treatment of ATTR amyloidosis. <sup>10</sup> Tafamidis binds to TTR at the thyroxine-binding site and inhibits TTR tetramer dissociation, the rate-limiting step in the amyloidogenic process. By stabilizing the tetrameric native state of TTR, tafamidis increases the activation barrier associated with tetramer dissociation and therefore mimics the tetrameric-stabilization effect observed with naturally occurring protective trans-suppressor variants. Tafamidis has been extensively studied for the treatment of ATTR amyloidosis in independent development programs in ATTR-PN and ATTR-CM.

Tafamidis meglumine 20 mg was the first disease-modifying therapy approved for the treatment of ATTR-PN and is currently labeled and approved for once-daily dosing for treatment of transthyretin amyloidosis in adult patients with stage 1 symptomatic polyneuropathy to delay peripheral neurologic impairment. Available in over 40 countries worldwide (excluding the United States) and marketed as VYNDAQEL, tafamidis meglumine 20 mg for treating ATTR-PN has demonstrated efficacy and safety and is backed

by a clinical development program including 1 controlled and 4 uncontrolled studies <sup>11-14</sup> The long-term effectiveness and safety of tafamidis in ATTR-PN has been further confirmed in real-world clinical practice, where it significantly delayed disease progression and improved overall quality of life. <sup>15-18</sup> As ATTR-PN is a progressive disease, early diagnosis and treatment are paramount, <sup>5</sup> although there are patients who continue to progress despite treatment. <sup>14,19</sup> In a real-world retrospective cohort study of 210 patients with hereditary ATTR amyloidosis treated with tafamidis meglumine 20 mg, tafamidis concentration (and consequently TTR kinetic stabilization) was identified as a predictor of response in a subset of patients, fueling the speculation that ATTR-PN patients might benefit clinically from a higher dose of. <sup>19</sup>

Tafamidis delivered as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily<sup>20</sup> was the first disease-modifying therapy approved for the treatment of cardiomyopathy of wild-type or hereditary transthyretin-mediated amyloidosis in adults to reduce cardiovascular mortality and cardiovascular-related hospitalization. Tafamidis is currently approved for the treatment of ATTR-CM in approximately 54 countries worldwide (including the United States). The efficacy and safety of tafamidis for treating ATTR-CM are supported by a clinical development program including one controlled and two uncontrolled studies in patients with ATTRv and ATTRwt cardiomyopathy. 21-23 The pivotal study of tafamidis in ATTR-CM, known as ATTR-ACT,<sup>23</sup> examined 20 mg and 80 mg (4 x 20 mg) of tafamidis meglumine with active dose groups pooled and compared with placebo for primary and secondary efficacy analyses. Both tafamidis doses significantly reduced the combination of all-cause mortality and cardiovascular-related hospitalizations over 30 months versus placebo. The individual 20-mg and 80-mg doses were further examined in post-hoc analyses of 30-month data from ATTR-ACT and interim data from the ongoing open-label long-term extension of ATTR-ACT.<sup>24</sup> After a median of 51 months' follow-up, patients initially treated with tafamidis 80 mg had a significant survival benefit compared with those initiated on the 20-mg dose. However, neurologic endpoints were not evaluated in the ATTR-CM development program, necessitating the use of alternative approaches to assess the potential benefit of tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily for delaying neurologic disease progression in ATTR amyloidosis.

Real-world data collection offers one such alternative. There are ATTRv-CM patients treated with tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, who are mixed phenotype and receiving cardiologic and neurologic assessments prior to and following treatment as part of standard clinical practice. This provides the opportunity to examine the effect of tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, on neurologic disease progression in these mixed-phenotype ATTRv-CM patients.

#### 8. RESEARCH QUESTION AND OBJECTIVES

## Primary Objective:

 To assess neurologic function before and after initiation of tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, in patients with mixed-phenotype ATTRv-CM in a real-world setting.

#### Secondary Objective:

 To assess mBMI in patients with mixed-phenotype ATTRv-CM receiving tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily, in a real-world setting.

#### 9. RESEARCH METHODS

## 9.1. Study Design

This will be an observational, retrospective cohort study using structured secondary anonymized data. Patients with mixed-phenotype ATTRv-CM receiving tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily for at least 6 months, will be identified. Relevant data will be extracted through at least 6 months following the initiation of tafamidis treatment.

Figure 9-1 Overview of Study Design



<sup>\*</sup>Charcot-Marie-Tooth neuropathy score v2 (CMTNS2); mBMI: Modified body mass index; MRC: Medical Research Council; NIS-CS: Neuropathy impairment score-composite score; NIS-LL: Neuropathy impairment score-lower limbs; PND: Polyneuropathy disability.

#### 9.2. Setting

The study will include patients with mixed-phenotype ATTRv-CM who are treated with tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily. All patients meeting the study enrollment criteria will be included.

#### 9.2.1. Inclusion Criteria

Patients must meet all the following inclusion criteria to be eligible for inclusion in the study:

- 1. Age ≥18 years at diagnosis.
- 2. Diagnosed with ATTRv-CM, mixed phenotype.
- 3. Treated with tafamidis (VYNDAQEL 80 mg [four 20-mg tafamidis meglumine capsules] orally once daily or VYNDAMAX 61 mg [one 61-mg tafamidis capsule] orally once daily) for ≥6 months.
- 4. Have had ≥1 pre- and ≥1 post-treatment neurologic assessments.\*

\*The pre-treatment neurological assessment will be at least 6 and up to 12 months prior to treatment initiation. The baseline assessment will be within 3 months before or 3 months after the start of tafamidis treatment. In the absence of baseline data within a+/-3 month window, structured data from exam notes may also be retrieved if available to align with real world practice. The post-treatment period will be at least 6months after treatment initiation.

Note: As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients is not required.

## 9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will be excluded from the study:

- 1. History of organ transplant.
- 2. Wild-type TTR genotype.
- 3. Individuals who are non-ambulatory.
- 4. Prior treatment with any disease-modifying therapy (investigational or approved) alone or in combination, except tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily.
- 5. Peripheral neuropathy attributed to causes other than ATTR amyloidosis (eg, diabetes mellitus, B12 deficiency, HIV infection).

## 9.3. Variables

## 9.3.1. Exposure Variables

Tafamidis treatment will be described using the variables in the table below.

**Table 9-1 Exposure Variables** 

| Variable | Role | Data source(s) | Operational Definition |
|---|---|---|---|
| Time to treatment initiation | Exposure | Research database | Calculated as time from ATTR-CM diagnosis to tafamidis initiation |
| Treatment start date | Exposure | Research database | Date of tafamidis treatment initiation |
| Treatment end date | Exposure | Research database | Date of end of tafamidis treatment |
| Treatment duration | Exposure | Research database | Calculated as time from treatment initiation to the end of treatment or last visit date |

## 9.3.2. Outcome Variable

For the primary and secondary objectives, the following clinical outcomes will be assessed. Neurologic progression scores are routinely collected in clinical practice.

**Table 9-2 Clinical Outcomes** 

| Variable | Role | Data source(s) | Operational Definition |
|---|---|---|---|
| Neurologic progression | | | |
| Neuropathy impairment<br>score– composite score<br>(NIS-CS) | Outcome | Research database | Data contains an assessment score for each muscle group or sensation area for motor strength/weakness, muscle stretch reflexes, and sensation. A final NIS-CS score will be calculated as a sum of these scores from the 3 sections ranging from 0 (normal) to 244 (total impairment). |
| Neuropathy impairment<br>score-lower limbs (NIS-<br>LL) | Outcome | Research database | Same as above, NIS-LL will be calculated using individual assessment scores for motor strength/weakness, muscle stretch reflexes and sensation, from lower body only, ranging 0 (normal) to 88 (total impairment). |
| Polyneuropathy disability<br>(PND) score | Outcome | Research database | A scoring system of the patient's walking capacity. It consists of four stages from stage 0 (no impairment) to stage IV (confined to a wheelchair or bedridden). |
| Medical Research Council<br>(MRC) Scale for Muscle<br>Strength | Outcome | Research database | The MRC scale of muscle strength uses a score of 0 to 5 to grade the power of a particular muscle group in relation to the movement of a single joint |
| Charcot-Marie-Tooth<br>neuropathy score v2<br>(CMTNS2) | Outcome | Research database | Composite of nine assessments: symptoms (three items), signs (four items), and neurophysiology (two items). It is designed to measure length-dependent |

## Tafamidis B3461099 NON-INTERVENTIONAL STUDY PROTOCOL Amendment 2, Version 3.0, 31 May 2023

| Variable | Role | Data source(s) | Operational Definition |
|---|---|---|---|
| | | | motor and sensory impairment in genetic neuropathies. Each assessment is scored on a $0-4$ point scale, reflecting severity of impairment. Patients are classified as mild (CMTNS $\leq 10$ ), moderate (CMTNS $11-20$ ), or severe (CMTNS $\geq 20$ ). |
| Overall health | | | |
| Height | Outcome | Research database | Height in centimeter or inches |
| Weight | Outcome | Research database | Weight in kilograms or pounds |
| Body mass index | Outcome | Research database | Recorded or calculated in kg/m <sup>2</sup> |
| Modified BMI (mBMI) | Outcome | Research database | Calculated as the product of BMI in kg/m <sup>2</sup> and serum albumin in g/L to compensate for peripheral edema. |

Patient demographic and clinical characteristics to be assessed are listed in Table 9-3.

Table 9-3 Patient Demographics, Clinical characteristics, and Comorbidities

| Variable | Role | Data source(s) | Operational Definition |
|---|---|---|---|
| Patient demographics | | | |
| Age | Baseline<br>characteristic | Research database | Patient age at baseline*; age groups will be determined by distribution of age. |
| Gender | Baseline<br>characteristic | Research database | Male/Female |
| Race | Baseline<br>characteristic | Research database | American Indian or Alaska<br>Native/Asian/Black or African<br>American/Native Hawaiian or Other<br>Pacific Islander/White |
| Ethnicity | Baseline<br>characteristic | Research database | Hispanic or Latino/Not Hispanic or<br>Latino |
| Clinical characteristics | | | |
| Age at ATTR-CM<br>diagnosis | Baseline<br>characteristic | Research database | Age at diagnosis in years |
| TTR genotype | Baseline<br>characteristic | Research database | Mutation in TTR gene associated with<br>ATTR amyloidosis (eg, Val122Ile,<br>Val30Met, Leu58His, Leu111Met) |
| Family history | Baseline<br>characteristic | Research database | No family<br>history/Parent/Siblings/Grandparent/<br>Other/Unknown |
| Comorbidities | | | |
| Charlson Comorbidity<br>Index (CCI)** | Baseline<br>characteristic | Research database | Based on comorbidities present at baseline*; grouped as 0, 1, 2, 3+ |

<sup>\*</sup>Baseline is defined as within 3 months prior to or 3 months following initiation of tafamidis. In the absence of baseline data within a +/- 3-month window, data outside this window may be used to align with real world practice.

#### 9.4. Data Source

The source of data for this study will be de-identified secondary data from an anonymized research database.

## 9.5. Study Size

No formal sample size calculation has been performed; all eligible patients treated at the study site will be included. It is estimated that at least 30 patients will be enrolled.

## 9.6. Data Management

Data will be transferred from the de-identified research database to OPEN Health's database server via encrypted external hard drive/disk or a secured file transfer protocol (FTP) server, which is locked in a secure room with physical access limited to server administrators. Network access to the database server will be restricted to the internet protocol (IP) addresses of project staff workstations on a limited access network behind a firewall system. Only

<sup>\*\*</sup>Individual comorbid conditions may be assessed based on feasibility assessment instead of CCI.

authorized personnel as indicated above will be provided with the password to use the media or log in to the server to access the data for analysis. The authorized personnel may download analytical datasets to their secured OPEN Health computers (encrypted and password protected). However, download to any personal computer will not be possible. Access to the received media and printed materials containing EMR data will be restricted to project staff and will be kept in a locked file cabinet. Aggregated analyses results will be presented at conferences and/or published in a journal with no patient-level data exposed.

The data will be used only for this specific study protocol. There will be no linkage of the data with any other data source. Patient IDs in the data are de-identified, and it will be impossible to trace patients' personal information (eg, name, mailing address) by using the patient ID. All analyses will be performed using Statistical Analysis System (SAS) version 9.4.

## 9.7. Data Analysis

Detailed methodology for summary and statistical analyses of data collected in this study will be documented in an SAP, which will be dated, filed, and maintained by the sponsor. The SAP may modify the plans outlined in the protocol; any major modifications of primary endpoint definitions or their analyses will be reflected in a protocol amendment.

## 9.8. Quality Control

To ensure programming quality and accuracy, the following steps will be taken:

- **Methodology review:** All methodology, from sample selection to variable calculation, will be discussed and reviewed at the time of project initiation.
- Operational definitions review: All operational definitions for calculated variables will be reviewed by the principal SAS programmer, a second SAS programmer, and Pfizer.
- Statistical review: The statistical methods utilized will be reviewed by a statistician
  as well as the SAS statistical programmer, project manager, senior scientific leader,
  and Pfizer.
- Output review: All SAS output will be initially reviewed by the SAS programmer for logic and reasonability. Output will then be reviewed by the project manager, senior scientific leader, and Pfizer. Additional reports will be run by the SAS programmer and Pfizer to ensure validation of SAS output.

During document preparation, quality control (QC) will include general proofreading and formatting, including but not limited to checks for errors related to spelling and grammar, font consistency, table/figure numbering, styles/header numbering, and general formatting/spacing. QC will also include confirming data (fact checking) and ensuring proper referencing, when applicable. For analyses and reports that utilize technical software, QC

will additionally include cross-checking internal methods/statistical review and ensuring clear presentation of findings. A corrective and preventative action plan will be part of analytic projects, with a documented deviation process and mechanisms in place to report serious deviations on the quality of/processes generating the data. The project officer or non-project senior staff member will serve as the internal resource for investigating and reporting serious deviations. The QC/quality assurance (QA) procedure will also be conducted for written communications, including meeting minutes and project-related emails, with internal team members and Pfizer.

#### 9.9. Limitations of the Research Methods

This study will have several limitations.

First, the retrospective and observational nature of our study may be subject to unmeasured confounding. However, a longitudinal before and after study design will be used to evaluate treatment effects in the same patient group. It will also be unlikely to have unmeasured time-varying patient factors since ATTR-CM is an inexorably progressive disease caused by genetic mutation or the aggregation of non-mutated, wild-type TTR due to aging. Study results could be affected by misclassification bias due to misreporting or misdiagnosis due to the similarity of ATTR-CM to other types of heart failure.

Second, the study will be limited to ATTRv-CM patients from a single center, potentially mitigating generalization of study results to other ATTRv-CM patient populations due to different patient characteristics or local practice patterns.

Finally, ATTR-CM is a rare disease. While the inclusion of <100 patients is generally considered a relatively small sample size, it is not for a rare disease. The sample size of the previous clinical trial that established the efficacy of once-daily tafamidis 20 mg on delaying neurologic progression in ATTR-PN was also relatively small given that this is a rare disease. <sup>11</sup> In addition, as the study will be exploratory in general, the sample size is not expected to be a limiting factor, and this will be taken into account when reporting the results.

#### 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient Information

This study will involve data that will exist in anonymized structured format and contain no personal patient information.

#### 10.2. Patient Consent

As this study will involve anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients will not be required.

## 10.3. Institutional Review Board (IRB)/Independent Ethics Committee

The study protocol will be submitted to the local IRB to apply for an exemption/waiver from IRB review prior to data transfer.

All correspondence with the local IRB will be retained and copies of correspondence filed in accordance with good pharmacoepidemiology practices (GPP).

#### 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor, and will follow generally accepted research practices described in Guidelines for GPP issued by the International Society for Pharmacoepidemiology, Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR), and United States Food and Drug Administration Guidance for Industry: Good Pharmacovigilance and Pharmacoepidemiologic Assessment.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start or a combination of existing structured data and unstructured data, which will be converted to structured form during the implementation of the protocol solely by a computer using automated/algorithmic methods, such as natural language processing. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results of this study will be made public by posting on clinicaltrials.gov. Further communication of these data may occur via abstracts and manuscripts.

#### 13. REFERENCES

- Ruberg FL, Grogan M, Hanna M, Kelly JW, Maurer MS. Transthyretin amyloid cardiomyopathy: JACC state-of-the-art review. *Journal of the American College of Cardiology*. 2019;73(22):2872-2891.
- 2. Ando Y, Coelho T, Berk JL, et al. Guideline of transthyretin-related hereditary amyloidosis for clinicians. *Orphanet journal of rare diseases*. 2013;8(1):1-18.
- 3. Mutations in Hereditary Amyloidosis. http://amyloidosismutations.com/attr.html. Accessed June, 29, 2021.
- 4. Conceição I, González Duarte A, Obici L, et al. "Red flag" symptom clusters in transthyretin familial amyloid polyneuropathy. *Journal of the Peripheral Nervous system*. 2016;21(1):5-9.
- 5. Conceição I, Damy T, Romero M, et al. Early diagnosis of ATTR amyloidosis through targeted follow-up of identified carriers of TTR gene mutations. *Amyloid*. 2019;26(1):3-9.
- 6. Maurer MS, Hanna M, Grogan M, et al. Genotype and phenotype of transthyretin cardiac amyloidosis: THAOS (Transthyretin Amyloid Outcome Survey). *Journal of the American College of Cardiology*. 2016;68(2):161-172.
- Castano A, Drachman BM, Judge D, Maurer MS. Natural history and therapy of TTRcardiac amyloidosis: emerging disease-modifying therapies from organ transplantation to stabilizer and silencer drugs. *Heart failure reviews*. 2015;20(2):163-178.
- 8. Rapezzi C, Quarta CC, Obici L, et al. Disease profile and differential diagnosis of hereditary transthyretin-related amyloidosis with exclusively cardiac phenotype: an Italian perspective. *European heart journal*. 2013;34(7):520-528.
- 9. Bulawa CE, Connelly S, DeVit M, et al. Tafamidis, a potent and selective transthyretin kinetic stabilizer that inhibits the amyloid cascade. *Proceedings of the National Academy of Sciences*. 2012;109(24):9629-9634.
- Burton A, Castaño A, Bruno M, et al. Drug Discovery and Development in Rare Diseases: Taking a Closer Look at the Tafamidis Story. *Drug Design, Development and Therapy*. 2021;15:1225.
- 11. Coelho T, Maia LF, da Silva AM, et al. Tafamidis for transthyretin familial amyloid polyneuropathy: a randomized, controlled trial. *Neurology*. 2012;79(8):785-792.
- 12. Coelho T, Maia LF, Da Silva AM, et al. Long-term effects of tafamidis for the treatment of transthyretin familial amyloid polyneuropathy. *Journal of neurology*. 2013;260(11):2802-2814.

- 13. Merlini G, Planté-Bordeneuve V, Judge DP, et al. Effects of tafamidis on transthyretin stabilization and clinical outcomes in patients with non-Val30Met transthyretin amyloidosis. *Journal of cardiovascular translational research*. 2013;6(6):1011-1020.
- Barroso FA, Judge DP, Ebede B, et al. Long-term safety and efficacy of tafamidis for the treatment of hereditary transthyretin amyloid polyneuropathy: results up to 6 years. *Amyloid*. 2017;24(3):194-204.
- 15. Lamb YN, Deeks ED. Tafamidis: a review in transthyretin amyloidosis with polyneuropathy. *Drugs*. 2019;79(8):863-874.
- Coelho T, Inês M, Conceição I, Soares M, de Carvalho M, Costa J. Natural history and survival in stage 1 Val30Met transthyretin familial amyloid polyneuropathy. *Neurology*. 2018;91(21):e1999-e2009.
- 17. Mundayat R, Stewart M, Alvir J, et al. Positive effectiveness of tafamidis in delaying disease progression in transthyretin familial amyloid polyneuropathy up to 2 years: an analysis from the transthyretin amyloidosis outcomes survey (THAOS). *Neurology and therapy*. 2018;7(1):87-101.
- 18. Huber P, Flynn A, Sultan MB, et al. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. *Amyloid*. 2019;26(4):203-209.
- 19. Monteiro C, Mesgazardeh JS, Anselmo J, et al. Predictive model of response to tafamidis in hereditary ATTR polyneuropathy. *JCI insight*. 2019;4(12)
- 20. Tafamidis label. https://www.fda.gov/media/126283/download. Accessed July 13, 2021.
- 21. Maurer MS, Elliott P, Merlini G, et al. Design and rationale of the phase 3 ATTR-ACT clinical trial (Tafamidis in Transthyretin Cardiomyopathy Clinical Trial). *Circulation: Heart Failure*. 2017;10(6):e003815.
- 22. Maurer MS, Grogan DR, Judge DP, et al. Tafamidis in transthyretin amyloid cardiomyopathy: effects on transthyretin stabilization and clinical outcomes. *Circulation: Heart Failure*. 2015;8(3):519-526.
- 23. Maurer MS, Schwartz JH, Gundapaneni B, et al. Tafamidis treatment for patients with transthyretin amyloid cardiomyopathy. *New England Journal of Medicine*. 2018;379(11):1007-1016.
- Damy T G-PP, Hanna M, Judge DP, Merlini G, Gundapaneni B, Patterson TA, Riley S, Schwartz JH, Sultan MB, Witteles R. Efficacy and safety of tafamidis doses in the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial (ATTR-ACT) and long-term extension study. *Eur J Heart Fail*. 2021;23(2):277-285.

## 14. LIST OF TABLES

Table 9-1 Exposure Variables

**Table 9-2 Clinical Outcomes** 

Table 9-3 Patient Demographics, Clinical characteristics, and Comorbidities

## 15. LIST OF FIGURES

Figure 9-1 Overview of Study Design

## ANNEX 1. LIST OF STAND ALONE DOCUMENTS

| Number | Document reference<br>number | Date | Title |
|---|---|---|---|
| 1 | Section 4 | 09 January<br>2023 | Real-World Effectiveness of Tafamidis<br>80 mg or 61 mg on Neurologic Disease<br>Progression in Patients with Mixed-<br>Phenotype ATTRv-CM |

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not required.

## ANNEX 3. ADDITIONAL INFORMATION

Not applicable.

## **Document Approval Record**

Document Name:

B3461099\_Non Interventional Protocol Amendment 2 version 3.0\_clea
n\_31May2023

B3461099\_Non Interventional Protocol Amendment 2 version 3.0\_clea
n\_31May2023

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 31-May-2023 20:55:31 | Final Approval |